CLINICAL TRIAL: NCT03140306
Title: Use of Low Dose CT Scanning of the Abdomen and Pelvis Using Model Based Iterative Reconstruction (MBIR) in Patients With Inflammatory Bowel Disease: Prospective Clinical Evaluation of Diagnostic Efficacy, Safety and Patient Outcome.
Brief Title: CT Using MBIR in Crohn's Disease: Prospective Clinical Evaluation of Diagnostic Efficacy, Safety and Patient Outcome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Owen O'Connor, Senior Lecturer, University College Cork
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MBIR study 2
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Radiology; Inflammatory Bowel Diseases
Keywords: Computed tomography; Model based iterative reconstruction; Low dose CT
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Split dose CT
Masking Description: the reader of the ct is blinded to the clinical presentation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose CT abdomen and pelvis (Experimental): Low dose computed tomography
  Interventions: Diagnostic Test: Patients who have had split dose CT
- Control dose CT abdomen and pelvis (Experimental): Control dose CT abdomen and pelvis
  Interventions: Diagnostic Test: Patients who have had split dose CT

INTERVENTIONS:
Diagnostic Test: Patients who have had split dose CT — Computed tomography

SUMMARY:
This study aims to assess the use of low dose CT reconstructed with MBIR for the assessment of patients with inflammatory bowel disease who need CT to assess for disease complications.

DETAILED DESCRIPTION:
The purpose of this study is to clinically validate the sole use of a low-dose computed tomography (CT) protocol to reduce the cumulative radiation dose in patients with inflammatory bowel disease. In an earlier study using the same CT parameters, the efficacy of the low dose technique was confirmed in the setting of a blinded retrospective review comparing the findings of the low dose and the conventional dose scan. The purpose of this study is to determine the reliability of the using low dose scan in a prospective clinical setting

This is to be achieved using Model Based Iterative Reconstruction (MBIR) which has been shown to result in diagnostically acceptable low-dose CT imaging while providing a significant reduction of ionising radiation dose to the patient. The authors aim to apply MBIR to their low dose protocol, and to facilitate diagnostic quality CT scanning of the abdomen and pelvis at an effective dose approximately four times less than what would normally occur with an abdominopelvic CT in patients with suspected active Crohn's disease (CD).

The authors plan to assess the diagnostic efficacy, safety and patient outcome of low dose CT reconstructed with MBIR in CD patients presenting to hospital with suspected acute mural and extramural complications.

Patients with inflammatory bowel disease referred to Cork University Hospital (CUH) will undergo two series of the abdomen and pelvis: a modified low dose protocol designed to impart a radiation exposure of 10-20% that of a routine abdominal and pelvic CT and a conventional dose protocol designed to impart an effective dose of 80-90% that of a routine abdominal and pelvic CT. Using this strategy, the image quality and diagnostic yield of the low dose CT can be compared with that of the conventional dose CT and no patient will incur additional radiation exposure as a result of recruitment into the study.

The low dose scan will be read alone initially by one of two experienced radiologists and the diagnostic report will come from this data set only. This report will be placed on the Picture Archiving and Communication System (PACS) to be used by the referring clinician who will then use the report/low dose scan images for patient management. This methodology is used to ascertain the clinical efficacy in a real world setting.

One month after the initial low dose read, the two Radiologists will read the conventional dose CT scans. Note will be made on the PACS report of either agreement or discrepancy with the original low dose report. Any important discrepancy will be highlighted to the referring clinician by either phone and/or a radiological alert email.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory bowel disease requiring CT to assess for disease complication

Exclusion Criteria:

* Pregnancy or children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Low-dose CT scanning of the abdomen and pelvis using Model Based Iterative Reconstruction (MBIR) in patients with inflammatory bowel disease: Clinical verification study | 2 years
  CT study assessing efficacy of reduced dose CT compared with normal dose CT

CONTACTS AND LOCATIONS:
Locations (1):
- Cork University Hospital, Cork, Co Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Grady J, Carey BW, Kavanagh RG, O'Connell A, O'Connor OJ, Kenny-Walsh E, Zulquernain SA, Maher MM, Shanahan F. Making computed tomography safer for patients with Crohn's disease. Scand J Gastroenterol. 2022 Feb;57(2):175-182. doi: 10.1080/00365521.2021.1994640. Epub 2021 Oct 26. PMID 34699288